CLINICAL TRIAL: NCT07126431
Title: Prospective Cohort Study on Refractory Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023089
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripehral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rheumatoid arthritis (RA) is a systemic autoimmune disease characterized by chronic erosive arthritis. Without timely and appropriate treatment, it can lead to joint destruction and disability. Current RA management emphasizes early diagnosis, early treatment, and a treat-to-target (T2T) approach to achieve disease remission as soon as possible.

In recent years, significant progress has been made in RA pharmacotherapy. With the clinical application of biologic disease-modifying antirheumatic drugs (bDMARDs) targeting cytokines and targeted synthetic DMARDs (tsDMARDs), treatment outcomes and prognosis have greatly improved. However, even with bDMARDs or tsDMARDs, some patients show poor response, maintaining moderate-to-high disease activity-a condition termed "refractory RA". Refractory RA has garnered increasing clinical attention, prompting the European Alliance of Associations for Rheumatology (EULAR) to establish a standardized definition and diagnostic criteria in 2020 to facilitate research.

Currently, effective treatments for refractory RA are lacking. These patients often present with extra-articular manifestations and comorbidities, posing significant therapeutic challenges. They exhibit higher rates of bone destruction and joint deformities, severely impairing work capacity and quality of life, thereby imposing heavy burdens on families and society.

Studies from Western countries estimate refractory RA prevalence at 5-20%, while its exact incidence in China remains unknown. Given regional disparities in rheumatology care and low overall RA remission rates in China, the proportion of refractory RA may be higher. Historically, this patient population has been understudied, and no prospective refractory RA cohort has been established in China.

Key factors contributing to refractory RA in China-including clinical phenotypes, immune subtypes, and predictive biomarkers-remain unclear. Developing personalized treatment strategies to manage refractory RA requires further exploration. There is an urgent need for prospective cohort studies to address these gaps.

This project aims to establish a dedicated refractory RA cohort to investigate its clinical and immune phenotypes under current T2T strategies and expanded bDMARD/tsDMARD insurance coverage. The investigators will explore potential clinical predictors and biomarkers, implement personalized therapies, and evaluate treatment efficacy, remission rates, and the predictive value of different phenotypes/subtypes. Additionally, the investigators will assess impacts on patient-reported outcomes (PROs) and quality of life. The findings will provide critical insights into refractory RA pathogenesis, predictive markers, and tailored therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 1987 American College of Rheumatology (ACR) classification criteria for RA or the 2010 ACR/European Alliance of Associations for Rheumatology (EULAR) classification criteria for RA.
2. Age >18 years.
3. Treatment with conventional synthetic DMARDs (csDMARDs) for at least 1 year.
4. Fulfill the EULAR definition of difficult-to-treat RA (refractory RA).
5. Provide written informed consent.

Exclusion Criteria:

1. Age <18 years.
2. Duration of DMARD therapy <1 year.
3. Patients unwilling to participate in the cohort study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis (RA) patients who are regularly followed up at the Department of Rheumatology and Immunology, Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DAS28-ESR | 2023-1-1 to 2025-12-31
  Disease Activity Score in 28 joints based on ESR

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China